CLINICAL TRIAL: NCT06449664
Title: ADT-Train - A New Training Concept for Men With Prostate Cancer Receiving Androgen Deprivation Therapy.
Brief Title: Training for Men Undergoing Androgen Deprivation Therapy.
Acronym: ADT-train
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Swedish School of Sport and Health Sciences (Other)
Collaborators: Norwegian School of Sport Sciences (Other); Karolinska Institutet (Other); Prostate Cancer Foundation (Other); Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-00964-01
Record Dates: First submitted 2024-04-04; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Prostate Cancer
Keywords: Androgen deprivation therapy (ADT); Flywheel training; High intensity training (HIT); Resistance training; Aerobic training
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): The participants will exercise twice weekly performing the newly developed training concept including flywheel resistance training followed by aerobic cycling intervals.
  Interventions: Behavioral: ADT-train
- Control group (No Intervention): The participants will receive usual care only.

INTERVENTIONS:
Behavioral: ADT-train — A new training concept is tested on men with prostate cancer receiving androgen deprivation therapy
  Arms: Exercise

SUMMARY:
The goal of this clinical trial is to evaluate the effects of a newly developed training concept on men with prostate cancer undergoing androgen deprivation therapy (ADT).

The main questions it aims to answer are:

* How feasible and safe is the new training concept?
* How efficient is the training concept to counteract side effects caused by ADT?

Researchers will compare the new training concept with usual care to evaluate how efficient the training concept is to counteract the ADT-related side effects.

Participants in the intervention group will perform the new training concept twice weekly for 12 weeks. Participants in the control group will only receive usual care. All participants will visit the laboratory at baseline and after 6 and 12 weeks to measure the primary and secondary outcomes.

DETAILED DESCRIPTION:
Detailed description of the training concept applied in the intervention:

The two weekly training sessions will be separated by at least two days and supervised by appropriately trained exercise professionals at The Swedish School of Sport and Health Sciences. The training includes a 10 min warm-up followed by 3-4 sets of 8 maximal repetitions on the flywheel machine followed by 16-24, 20 s intervals on a Monark cycle ergometer. The intervals will be performed as 3 blocks with the intention to execute 8 intervals in each block. When a participant manages to perform all 3 blocks with 8 intervals in each block (a total of 24 intervals) the resistance will be increased by ~20 W. The rest period between the intervals will be set to 10 s and the rest between the blocks to 2 min. The starting workload of the intervals will be individually adjusted to ~115 % of the participant's power output at VO2peak. The total duration of a training session will be 30-40 min (including worm-up).

ELIGIBILITY:
Inclusion Criteria:

1. signed informed consent
2. histologically confirmed localised or locally advanced prostate cancer
3. planned radiotherapy in combination with ADT for at least six months (unfavorable intermediate risk and high-risk prostate cancer) with curative intent and with no known metastasis.

Exclusion Criteria:

1. very high risk localised prostate cancer planned for radiotherapy and ADT plus abiraterone and cortisone
2. localized prostate cancer planned for radiotherapy without ADT
3. on-going or previously treated with ADT or other hormonal treatments
4. have any contraindications to physical testing/exercise as per the ACSM guidelines
5. unable to comply with study procedures

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12-20 (Estimated)

PRIMARY OUTCOMES:
Aerobic fitness | Baseline and after 6 and 12 weeks
  VO2peak (ml/kg/min); incremental ramp test on a cycle ergometer
Maximal leg strength | Baseline and after 6 and 12 weeks
  Isometric squat test (N) measured on force plates

SECONDARY OUTCOMES:
Body fat | Baseline and after 6 and 12 weeks
  Assessed by dual-energy x-ray absorptiometry (DEXA) (kg)
Lean body mass | Baseline and after 6 and 12 weeks
  Assessed by dual-energy x-ray absorptiometry (DEXA) (kg)
Bone mineral density | Baseline and after 6 and 12 weeks
  Assessed by dual-energy x-ray absorptiometry (DEXA) (g/cm2)
Quadriceps cross-sectional area | Baseline and after 6 and 12 weeks
  Assessed by ultrasound (mm)
Static balance | Baseline and after 6 and 12 weeks
  One leg balance test on the right and the left foot. Time to first footing is measured and the number of footings during 60s.
Walk capacity | Baseline and after 6 and 12 weeks
  Usual and fast pace 6m walk test (s)
Lower body muscular endurance | Baseline and after 6 and 12 weeks
  30 s chair stand test. Maximal number of sit-to-stand repetitions during 30 s.
Blood pressure | Baseline and after 6 and 12 weeks
  Assessed by an automated blood pressure monitor (mmHg).
Whole body glucose uptake | Baseline and after 6 and 12 weeks
  Assessed by an oral glucose tolerance test in which the participants will ingest a standardized glucose drink and blood glucose levels will be monitored throughout a period of 2 hours (mmol/L).
Whole body insulin response | Baseline and after 6 and 12 weeks
  Assessed by an oral glucose tolerance test in which the participants will ingest a standardized glucose drink and blood insulin levels will be monitored throughout a period of 2 hours (μU/mL).
Blood biomarkers related to cardiovascular disease. | Baseline and after 6 and 12 weeks
  Assessed by high-multiplex immunoassays quantifying proteins associated with biological functions linked to cardiovascular diseases. Approximately 100 proteins will be assessed. Examples of proteins are: C-Reactive Protein (CRP), Tissue Factor (F3), and Thrombomodulin (THBD).
Muscle fiber cross-sectional area (CSA) | Baseline and after 12 weeks
  Type I and type II muscle CSA will be assessed by immunohistochemistry (µm2).
Muscle fiber distribution | Baseline and after 12 weeks
  Type I and type II muscle fiber distribution will be assessed by immunohistochemistry (%).
Capillary content | Baseline and after 12 weeks
  The number of capillaries per muscle fiber will be assessed by immunohistochemistry.
Myonuclei content | Baseline and after 12 weeks
  The number of myonuclei per muscle fiber CSA will be assessed by immunohistochemistry.
Satellite cell content | Baseline and after 12 weeks
  The number of satellite cells per muscle fiber CSA will be assessed by immunohistochemistry.
Mitochondrial content | Baseline and after 12 weeks
  Mitochondrial content will be assessed by measuring citrate synthase activity in homogenized muscle samples (mmol/kg/dw/min).
Mitochondrial respiration | Baseline and after 12 weeks
  Mitochondrial respiration will be assessed by respirometry of permeabilized muscle fibers (respiration ratio).
Genome-wide DNA methylation | Baseline and after 12 weeks
  Assessed by Illumina EPIC arrays to identify epigenetically regulated genes and pathways associated with exercise and the ADT-treatment.
Transcriptome-wide RNA expression | Baseline and after 12 weeks
  Assessed by RNA-sequencing to identify differently regulated genes and pathways associated with exercise and the ADT-treatment.
Protein expression | Baseline and after 12 weeks
  Assessed by Western Blot and ELISA (AU). This could for example be proteins related to genes identified by the genome-wide DNA methylation analysis or transcriptome-wide RNA expression analysis.
Gene expression | Baseline and after 12 weeks
  Assessed by quantitative real-time PCR (AU). This could for example be genes identified by the genome-wide DNA methylation analysis or transcriptome-wide RNA expression analysis.
Cancer treatment-related symptoms | Baseline and after 6 and 12 weeks
  Assessed by the National Prostate Cancer Register (NPCR) form. Scores scaled from 0 to 7. A higher score indicates more severe symptoms.
Physical activity | Baseline and after 6 and 12 weeks
  Assessed by the physical activity questionnaire. Scores scaled from 1 to 8. A higher score indicates a more physically active participant.
Physical and psychological health | Baseline and after 6 and 12 weeks
  Assessed by the Short Form Health Survey (SF-36). Scores scaled from 1 to 6. A higher score indicates better physical and psychological health.
Anxiety and depression | Baseline and after 6 and 12 weeks
  Assessed by the Hospital Anxiety and Depression Scale (HADS). Scores scaled from 0 to 3. A higher score indicates more anxiety and depression.
Cancer and treatment-related fatigue | Baseline and after 6 and 12 weeks
  Assessed by the Multidimensional Fatigue Inventory survey (MFI-20). Scores scaled from 1 to 5. A higher score indicates more fatigue.

CONTACTS AND LOCATIONS:
Locations (1):
- Swedish School of Sport and Health Sciences, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided